CLINICAL TRIAL: NCT01639638
Title: Randomised, Blind and Placebo-controlled Trial for the CIGB-300 Perilesional Application in Two Dose Levels in the Recurrent and Non Recurrent Genital Condyloma
Brief Title: Recurrent and Nonrecurrent Condyloma Treatment
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CONDI 02 AR
Record Dates: First submitted 2012-05-14; First posted 2012-07-13 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Recurrent Condyloma; Nonrecurrent Condyloma
Keywords: Recurrent and non-recurrent genital condyloma
MeSH Terms: conditions — Condylomata Acuminata; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: PROAPOPTOTIC PEPTIDE CIGB 300
- CIGB-300 - 5 mg (Experimental)
  Interventions: Drug: PROAPOPTOTIC PEPTIDE CIGB 300
- CIGB-300 - 15 mg (Experimental)
  Interventions: Drug: PROAPOPTOTIC PEPTIDE CIGB 300

INTERVENTIONS:
Drug: PROAPOPTOTIC PEPTIDE CIGB 300 — CIGB 300,in INTRALESIONAL on day 3 of each 48 HOURS.

SUMMARY:
Treatment is considered successful if the difference in the response in the reduction of the affected area is above 30% for any of the doses compared to placebo Patients will be randomised to 1 of 3 treatment arms

1. Placebo
2. CIGB-300 - 5 mg
3. CIGB-300 - 15 mg

A two week screening visit will take place to assess patient eligibility, at least 2 to 5 target lesions (area of the lesion between 20 to 80 mm2), should be identified. Patients included in the study will be randomly assigned to one of three study arms. Treatment consists of 3 perilesional applications at the base of the target lesion every 48 hours with a window of ±24hs.

After each application the potential local and systemic adverse events will be identified and monitored.

After the last application is made, weekly clinical evaluations for 3 weeks and then every two weeks, until week 12 will take place. At this time, clinical assessment of efficacy will be carried out that will define the response to treatment.

After this visit, patients will be followed every 3 months until one year after the last treatment has been completed to confirm response and long-term security of the CIGB-300 application.

At screening, at 2 and 8 weeks as well as at 6 and 12 months post-treatment blood studies will be conducted to assess the safety from the systemic point of view.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the patient
2. Women with clinical diagnosis of recurrent and non recurrent genital condyloma
3. Presence of a condylomatous lesion or area of external confluent condylomatous lesions of not less than 20 or more than 80 mm2
4. The number of warts should be between 2 and 20
5. External genital warts or in perigenital regions
6. Negative pregnancy test
7. Age between 18 and 65 years inclusive

Exclusion Criteria:

1. Having received surgery treatment, ablative or immunomodulator treatment during the 30 days prior to inclusion
2. Presence of genital warts only located in the cervix, vagina, bladder or rectum
3. Pregnancy and lactation
4. Patients of childbearing age who are not using an adequate contraception method during treatment to prevent pregnancy.
5. Inadequately controlled chronic diseases (hypertension, diabetes, chronic kidney failure, heart failure, hyperthyroidism, malignant neoplasms, epilepsy, severe mental depression)
6. Patients with previous diagnosis of bleeding disorders and other chronic blood disorders (von Willebrand disease, haemophilia, leukaemia) or use of anticoagulants within 30 days before the study
7. Current genital herpes, which requires application of topical antivirals
8. Immunosuppressive disease, current intake of immunosuppressive/ immunomodulatory drugs within 30 days before the study.
9. Autoimmune Diseases (Lupus Erythematosus, Rheumatoid Arthritis, Multiple Sclerosis, Diabetes)
10. Severe allergy history as urticaria, dermatitis or persistent bronchitis and bronchial asthma
11. Febrile illness (temperature greater than 38ºC) at the time or within 24 hours prior to administration of the product or suspected acute infectious disease by clinical examination
12. Diseases that compromise the patient's consciousness or the ability to give informed consent or to collaborate in the study
13. Concomitant skin lesions that prevent the administration of condylomatous lesions at the proposed site
14. Participating in another clinical trial

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete response of target lesion in each study group | Up to one year
Number of patients with adverse events during the application of the study drug | Up to one year

SECONDARY OUTCOMES:
Effect of the perilesional application of CIGB300 in the reduction in the number and area of genital warts lesions treated directly | Up to one year
Locoregional effect of CIGB300 by assessing the area and number of genital warts lesions not directly treated | Up to one year
Effect of CIGB300 to avoid recurrence of the lesions | Up to one year
Optimal dose, in comparison with placebo | Up to one year
Number of patients with adverse events | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio Elea SACIFyA, Capital Federal, Buenos Aires, Argentina

REFERENCES:
- See also: Related Info — http://www.elea.com